CLINICAL TRIAL: NCT00926874
Title: A Comparative Study of Structural and Functional Arterial Properties After an Ischaemic Stroke or an Acute Coronary Syndrome
Brief Title: Comparative Study of Arterial Properties After an Ischaemic Stroke or an Acute Coronary Syndrome
Acronym: AVC/SCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: University Hospital, Grenoble, Pr Jean-PHilippe BAGUET
Other Study IDs: 0401; DGS 2008/0443
Record Dates: First submitted 2009-03-23; First posted 2009-06-24 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Ischemic Stroke; Acute Coronary Syndrome; Obstructive Sleep Apnea Syndrome
Keywords: ischaemic stroke; acute coronary syndrome; obstructive sleep apnea syndrome; brachial endothelial function; blood pressure; aortic stiffness
MeSH Terms: conditions — Ischemic Stroke; Acute Coronary Syndrome; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients who presented an ischaemic stroke(full stroke or TIA)
- 2: patients who present an acute coronary syndrome (ACS).

SUMMARY:
A pilot, prospective, comparative study. To include both male and female patients who have presented an ischaemic stroke (full stroke or TIA) or an ACS, 5 to 30 days prior to inclusion.

The proposed study aims to investigate and analyse the differences in functional and structural arterial properties between the patients who presented an ischaemic stroke and those who presented ACS. The hypothesis is that the patients in both groups will present differences partly in terms of their "traditional" cardiovascular risk factors, but also in terms of their arterial properties. All of the confounding factors studied (cardiovascular risk factors, treatments) will be taken into account in order to explain the differences in the arterial properties found between the two groups. Furthermore, the prevalence of signs and symptoms in the two populations will be studied.

DETAILED DESCRIPTION:
A comparative study of structural and functional arterial properties after an ischaemic stroke or an acute coronary syndrome

Objectives:

Primary:

* To determine whether there is a difference in the biomechanical properties of the carotid arteries, assessed by studying their stiffness, after an acute vascular event, depending on whether the event is an ischaemic stroke (either a full stroke or a transitory ischaemic attack (TIA)) or an acute coronary syndrome (ACS).

Secondary:

* To determine whether there is a difference in aortic stiffness and brachial endothelial function after an acute vascular event, depending on whether the event is an ischaemic stroke (full stroke or TIA) or an ACS.
* To compare the blood pressure (BP) levels and the vascular parameters of the two patient groups (the ischaemic stroke group and the ACS group).
* To determine whether there is a difference between the respiratory parameters recorded during sleep after an acute vascular event, depending on whether the event is an ischaemic stroke (full stroke or TIA) or an ACS.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Between 40 and 70 years of age
* Who have given their written consent
* Who have presented the following between 5 and 30 days prior to inclusion:
* either an ischaemic stroke (full stroke or TIA) that has been stabilised from a neurological point of view, with no haemorrhage but with direct signs of ischaemia on the cerebral imaging (computed tomography or MRI), diagnosed during patient questioning and/or the clinical examination;
* or an ACS that has been stabilised from a cardiological point of view, with troponin elevation in at least 2 samples and/or ECG changes that indicate acute myocardial ischaemia, diagnosed during patient questioning.
* Who are affiliated to the French social security system

Exclusion Criteria:

* For patients included in the ACS group

  * Stroke less than 6 months ago
  * Coronary bypass between the start of their hospitalisation for ACS and inclusion
* For patients included in the stroke group

  * Emboligenic heart disease
  * ACS less than 6 months ago
* For all patients

  * Atrial fibrillation or flutter, or frequent extrasystole (more than 10/minute) upon inclusion
  * History of surgery or carotid stenting
  * Very reduced mobility meaning that they cannot remain standing without assistance or without using a walking stick

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented an acute vascular event :an ischaemic stroke (either a full stroke or a transitory ischaemic attack (TIA)) or an acute coronary syndrome (ACS).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2005-11; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
biomechanical properties of the carotid arteries | 1-6 months

SECONDARY OUTCOMES:
aortic stiffness and brachial endothelial function | 1-6 months
blood pressure (BP) levels and the vascular parameters | 1-6 months
respiratory parameters recorded during sleep | 1-6 months

CONTACTS AND LOCATIONS:
Overall Officials: BAGUET Jean Philippe, Professor, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France

REFERENCES:
- [Derived] Barone-Rochette G, Vanzetto G, Detante O, Quesada JL, Hommel M, Mallion JM, Baguet JP. Imaging of functional and structural alterations of large arteries after acute ischaemic atherothrombotic stroke or acute coronary syndromes. Arch Cardiovasc Dis. 2014 Aug-Sep;107(8-9):443-51. doi: 10.1016/j.acvd.2014.05.007. Epub 2014 Jul 10. PMID 25023004